CLINICAL TRIAL: NCT02361229
Title: Skin Cancer in Swiss Transplant Cohort Study
Acronym: SCSTCS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2014-0276
Record Dates: First submitted 2015-02-05; First posted 2015-02-11 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
It's known that organ transplant recipients with long-term drug-induced immunosuppression have a increase of the life-time incidence of squamous cell carcinoma. This study will analyze the incidence and type of skin cancer in the Swiss Transplant Cohort Study and the association with exposure to immunosuppressive and antiinfective drugs and other parameters like age or gender of organ transplant recipients.

DETAILED DESCRIPTION:
Organ transplant recipients with long-term drug-induced immunosuppression have an increase of the life-time incidence of squamous cell carcinoma and are also affected at an earlier age than the general population. In organ transplant recipients prognosis of squamous cell carcinoma differs due to more rapid growth, less differentiation and higher risk for metastases in comparison to the general population. Epidemiological data indicate that the risk of skin neoplasms in organ transplant recipients is related to the cumulative exposure to immunosuppressive drugs over time. It remains unclear wether this risk differs between drug classes.

This study is a prospective observational cohort study of kidney, heart, lung, liver, pancreas and small bowel transplant recipients enrolled into the Swiss Transplant Cohort Study (STCS).

Since 2008 almost all organ transplant recipients in Switzerland are enrolled to the STCS. The STCS collects

* baseline patient and case data: date of transplantation, age, gender, type of transplanted organ, past immunosuppression
* follow-up patient and case data: organ rejection with type and date of rejection, type of immunosuppression in response to organ rejection, graft loss with date of graft loss, immunosuppressive drug treatment, other drug treatment, death, drop out, occurrence of cancer and infections)
* drug exposure data (with start and stop dates): induction immunosuppressive drugs (Basiliximab, Rituximab, Thymoglobulin, ATG, ATGAM, IG iv, Plasmapheresis), maintenance immunosuppressive drugs (Cyclosporine A, Glucocorticoids, Tacrolimus, Mycophenolate mofetil, Everolimus, Azathioprine, Sirolimus, EC-MPA), infectious disease prophylaxis (e.g. TM-Sulfamethoxazole, Valaciclovir, Fluconazole, Atovaquone, Voriconazole, Quinolone), other drugs (e.g. Statins, beta-Blockers, oral antidiabetics).

The investigators will statistically illustrate the incidence, prevalence and type of skin neoplasms in the STCS. The investigators will show the association of the incidence of skin neoplasms and the exposure to different immunosuppressive drugs, other drugs and other parameters in the STCS (e.g. age, gender).

ELIGIBILITY:
Inclusion Criteria:

* solid organ transplant recipients within the STCS
* patients with multiple organ transplantations will be included as well
* patients within the STCS, who gave the informed consent to use their data
* patients with graft loss will remain in the study, since they remain at risk of skin cancer development

Exclusion Criteria:

* organ transplant recipients of non-solid organs (e.g. hematopoetic stem cell transplantation) within the STCS

Min Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Solid organ transplant recipients within the STCS.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Skin Cancer in SOTRs | 10 years
  skin cancer event
Incidence and type of skin neoplasms in STORs | 10 years
  skin neoplasm event

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, Prof MD, Principal Investigator — University Hospital Zurich, Dermatology
Locations (1):
- University Hospital Zurich, Dermatology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Share data with Swiss Transplant Cohort Study. Future projects can obtain data after project request is approved.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2019-2080
Access Criteria: STCS scientific committee approval and ethical committee approval (IRB)